CLINICAL TRIAL: NCT02774304
Title: Assessment of Arterial Dynamic Elastance as a Function Variable of Arterial Load, Derived From Both Non-invasive and Invasive Haemodynamic Variables.
Brief Title: Assessment of Arterial Dynamic Elastance as a Function Variable of Arterial Load
Acronym: Eadyn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Eadyn version 1.0
Record Dates: First submitted 2016-04-01; First posted 2016-05-17 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hypovolemia
Keywords: elastance; fluid responsiveness
MeSH Terms: conditions — Hypovolemia | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arterial line (Active Comparator): invasive haemodynamic monitoring
  Interventions: Device: arterial line; Device: Cheetah®
- Cheetah® (Experimental): non-invasive cardiac output
  Interventions: Device: arterial line; Device: Cheetah®

INTERVENTIONS:
Device: arterial line — In mechanically ventilated patients systolic pressure variation will be captured and passive leg raising with positive result fluid filling will be initiated.
Device: Cheetah® — In mechanically ventilated patients systolic pressure variation will be captured and passive leg raising with positive result fluid filling will be initiated.

SUMMARY:
The goal of the study is to determine Eadyn as a functional measure of arterial load, in conjunction with other actual afterload indices, derived from both invasive arterial pressure tracing and non-invasive signals, such as arterial saturation, non-invasive cardiac output obtained by bio-reactance, and non-invasive stroke volume. A secondary aim is the correlation of the different non-invasive signals with the invasive arterial pressure tracing characteristics.

DETAILED DESCRIPTION:
Fifteen patients, who provide written informed consent, will be included. All of them are scheduled for a major surgical intervention, in whom standard haemodynamic monitoring includes arterial pressure monitoring.

Non-invasive wired patches, connected to a Cheetah cardiac output monitor, will be installed, as well as traditional haemodynamic monitoring (ECG, SaO2, non-invasive blood pressure). A computer link between a Philips monitor (MP50 or MP70) is made, to obtain selected curves in a digital format for post-intervention processing. After awake insertion of an arterial catheter in the radial or brachial artery and induction of anaesthesia, patient becomes intubated and mechanically ventilated.

Before surgery, following data will be registered for 5 min.: ECG, invasive arterial pressure tracing, cardiac output (Cheetah monitor), SaO2 tracing, arterial pressure tracing and pulse pressure and stroke volume variation (Nexfin).

When SVV > 15%, the operation table will be put in Passive Leg Raising (PLR) to optimize the filling status of the patient (test of preload dependency). When positive haemodynamic reaction is present, the patients will obtain a rapid infusion bolus of 250 ml of crystalloids.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for a major surgical intervention, in whom standard haemodynamic monitoring includes arterial pressure monitoring.

Exclusion Criteria:

* Minor surgery and absence of arterial pressure monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Dynamic Elastance | 2 minutes
  determination of stroke volume and pulse pressure variation: ratio of SPV/SVV

SECONDARY OUTCOMES:
Stroke volume variation (SVV) | 2 minutes
  Variation of stroke volume (area under the arterial or oxygen saturation curve) during mechanical ventilation
Systolic pressure variation (SPV) | 2 minutes
  Variation of systolic pressure or peak oxygen saturation during mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Michel Vervoort, Ir, Study Director — Universitair Ziekenhuis Brussel; Jan Poelaert, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Tina Maes, MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No